CLINICAL TRIAL: NCT02462642
Title: Chronic Effect of Brahmi on Cognition Performance and Anxiety in Healthy Indian Adults and Exploration of Pharmacokinetic Properties of Brahmi Components in Healthy Adult Males.
Brief Title: Effect of Bacopa Monniera Extract on Cognition and Anxiety and Exploration of PK Properties
Acronym: Yaaddasht
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 08068B
Record Dates: First submitted 2014-09-16; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Cognition; Anxiety; Pharmacokinetics
Keywords: Brahmi, Cognition, Anxiety, Pharmacokinetics
MeSH Terms: conditions — Anxiety Disorders | interventions — Centella asiatica extract; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Brahmi - 36 subjects (Experimental): 36 subjects both male and female will consume 2 capsules of Brahmi for 84 days.
  Interventions: Dietary Supplement: Brahmi
- Placebo- 36 subjects (Placebo Comparator): 36 subjects male and female who will take 2 capsules of placebo every day
  Interventions: Other: Placebo
- Brahmi - 8 Subjects (Experimental): For PK part of the study 8 male subjects will be taken for treatment arm. Each volunteer will consume 2 capsules of Brahmi each day for 84 days.
  Interventions: Dietary Supplement: Brahmi
- Placebo- 4 subjects (Placebo Comparator): 4 male subjects in PK part will be in the placebo arm. Each volunteer will consume 2 capsules of Brahmi each day for 84 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Brahmi — Brahmi extract - 225 mg filled in each hard gelatin capsule. Two such capsules per day, to be taken by the subjects for 12 weeks.
  Other Names: Bacopa monniera
  Arms: Brahmi - 36 subjects
Other: Placebo — Dry maize starch filled in identical hear gelatin capsule. Two such capsules will be taken by each subject per day for 12 weeks.
  Other Names: Dry Starch
  Arms: Placebo- 36 subjects
Dietary Supplement: Brahmi — Brahmi Extract 225 mg filled in hard gelatin capsule. Two such capsules will be consumed by the subjects each day for 84 days.
  Other Names: Bacopa monniera
  Arms: Brahmi - 8 Subjects
Other: Placebo — Placebo capsules - Dry starch filled in identical hard gelatin capsules
  Other Names: Maize Starch capsules
  Arms: Placebo- 4 subjects

SUMMARY:
The Indian Ayurvedic herb Brahmi (Bacopa monniera) has been used to improve cognitive functions in Indian sub-continent for many years and previous intervention studies have shown positive effects of Brahmi on cognitive performance in adults. However, the studies are conducted on various fractions and extracts and there is high likelihood of variability of composition amongst the fractions/extracts tested in these studies. Furthermore, although the findings of the previous studies overlap to some extent, they are not consistent and there is a need to replicate these findings.

Further, even though Brahmi has been studied for its chemical composition and its therapeutic benefits as a whole, there are still severe gaps with respect to the complete composition of the Brahmi plant or its extracts. No published data exist on the Pharmacokinetics (PK) properties of Brahmi components. Hitherto, the evidence and the mechanistic details are still speculative and the biological activity is still phenomenological. Because of this severe knowledge gap, this study will try to repeat the findings on cognitive performance and at the same time also explore the plasma levels of its components in order to initiate the understanding of ADME aspects and its linkages to the biological effect.

DETAILED DESCRIPTION:
The study is proposed to be a randomised, double blind, placebo-controlled study with parallel groups. The duration of the study will be 12 weeks.

For cognition and Anxiety part, each selected subject will be paying 4 visits to clinical site for the whole study. Screening/selection will be done on visit 1, baseline on visit 2 and post-intervention assessment on visit 3. Subjects will be asked to appear for an interview before the investigators once more within one month of completion of intervention to take care of issues, if any. This will be 4th and last visit.

Each subject will be assessed at baseline (Week 1, Day 1); while post intervention assessment will be carried out immediately on the completion of the 12 weeks. Considering the 84 days duration of the study, + 3 days for the intervention period will be acceptable. The exact intervention duration will be documented in days for each subject.

On each of the two measurement days (baseline and post intervention), the same test battery will be administered by the same examiner. The outcome measures of this battery include Verbal Learning and Memory, Information Processing, Attention and Interference and Anxiety. The test battery will be administered in English.

On each of the measurement day the subject will spend a maximum of 1½ hours at the clinical site. Subjects will be examined in the morning at approximately the same time during both measurement days to keep conditions constant across the subjects and for baseline and post intervention assessments.

Each subject participating in Pharmacokinetics (PK) part, will pay 6 visits. Visit 1 will be screening, Visit 2,3 and 4 for initial blood withdrawal and visit 5 will post intervention blood sampling. Subjects will be asked to appear for an interview before the investigators once more within one month of completion of intervention to take care of issues, if any, which will be visit 6.

Blood sampling will be done at 0,1,2,4,8,24,48 hours and one sample at the endo of 12 weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects in the age between 35 and 60 at start of the study
* BMI BETWEEN 20 and 30 kg/m2
* Apparently mentally and physically healthy
* Willing to refrain from foods and supplements that contain caffeine, such as coffee, tea, chocolate, cola and energy drinks from 9 PM on the evening before each test day.
* Willing to refrain from supplements that are likely to have an effect on cognitive performance
* Having Haemoglobin counts more than 11 mg/ DL and normal blood profile in Physician's opinion (only for pharmacokinetic part)

Exclusion Criteria:

* Being on a medically prescribed- or slimming diet
* Reported weight loss/gain > 10% of body weight in the 6 month preceding pre-study examination
* Using herbal supplements or dietary supplements meant for improving cognitive performance
* Undergoing medical treatment that may interfere with the study outcome
* Using systemic antibiotics in the period of 3 months prior to or during the run-in period of the study
* Scoring above the cut off 9 on the GHQ28
* Pregnancy during the study period or in the six months prior to pre-study investigation
* Reported lactating 6 weeks before pre-study investigation and during the study
* Intense exercise >10 h/w
* Being colour-blind or dyslexic
* Hearing or vision impairments
* High alcohol consumption as indicated by a score of 4 or more on the AUDIT-C
* Smoking and/ or chewing tobacco during the past 6 months
* Recreational drug use during the past 6 months

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in Delayed recall from Baseline at day 0 to post intervention at day 84 | "0" (baseline) day and "84" day (Post Intervention)
  Rey Auditory Verbal Learning Test, Delayed recall

SECONDARY OUTCOMES:
Total learning, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Rey Auditory Verbal Learning Test, total learning,
Pro-active interference, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Rey Auditory Verbal Learning Test, pro-active interference
Retro-active interference, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Rey Auditory Verbal Learning Test, retro-active interference
Inspection Time, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Inspection Time Task: Inspection Time
Reaction time, correct responses, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Rapid Visual Information Processing Test, reaction time, correct responses
Reaction time, errors, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Rapid Visual Information Processing Test, reaction time, errors
Interference, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  Stroop Task, Interference
State, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  State-trait Anxiety Inventory, state
Trait, change between baseline at day 0 to post intervention at day 84 | "0" day and "84" day
  State-trait Anxiety Inventory, trait
Absorption constant | "0" day and "84" day
  Constant of absorption of the Brahmi components
Tmax | "0" day and "84" day
  Time of highest concentration in blood of the Brahmi components
T1/2 | "0" day and "84" day
  Half-life of the of the Brahmi components
Metabolites | "0" day and "84" day
  Scan for potential metabolites of the Brahmi components

CONTACTS AND LOCATIONS:
Overall Officials: Krishnamachari Srinivasan, Principal Investigator — St. John's Research Institute
Locations (1):
- St Johns Research Institute, Bangalore, Karnataka, India